CLINICAL TRIAL: NCT00866476
Title: Safety, Immunogenicity, and Efficacy Following Experimental Challenge of CVD 1208S, a Delta guaBA, Delta Sen, Delta Set Shigella Flexneri 2a Live, Oral Vaccine: Phase IIa Vaccination Study
Brief Title: Safety and Efficacy Study of CVD 1208S, a Live, Attenuated Oral Vaccine to Prevent Shigella Infection: Phase IIa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reactogenicity met study halting criteria
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: PATH (Other)
Responsible Party: Principal Investigator, Karen Kotloff, Professor of Pediatrics and Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00040710 Phase IIa; Shigella CVD 27000 (Other: University of Maryland Center for Vaccine Development)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Shigella
Keywords: Shigella; Vaccine; Mucosal immunity
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine-recipients (Experimental)
  Interventions: Biological: CVD 1208S, a Shigella flexneri 2a live, oral vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CVD 1208S, a Shigella flexneri 2a live, oral vaccine — CVD 1208S consists of freshly harvested ∆guaBA, ∆sen, ∆set S. flexneri 2a strain 2457T suspended in phosphate buffered saline to reach the desired inoculum Form: liquid Dose: 10 to the 9th power CFU in 1.0 ml Route: oral.
  Arms: Vaccine-recipients
Other: Placebo — 30 ml of buffer solution (2.0 grams of NaHCO3 dissolved in 150 ml of sterile water) without bacteria, to which food grade corn starch, USP is added, as necessary, to match the turbidity of the vaccine inoculum
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CVD 1208S (a live, attenuated, oral vaccine) is safe and effective in the prevention of Shigella infection.

DETAILED DESCRIPTION:
The study comprises a Phase 2 vaccination study and a Phase 2b challenge study. The primary objectives of the Phase 2 vaccination study are: 1. To evaluate, in healthy volunteers, the safety and clinical acceptability of three spaced doses (one month apart) of an investigational, live, oral, attenuated vaccine called CVD 1208S, with particular attention to the occurence of diarrhea, dysentery, and fever, and 2. To characterize immune responses following ingestion of this vaccine. The primary objective of the Phase 2b challenge study is to measure the protective efficacy of 3 spaced doses of vaccine after ingestion of an oral challenge strain called Shigella flexneri 2a strain 2457T.

Shigella is a leading cause of disease and death among children younger than 5 years living in developing countries. The difficulty controlling this infection has led experts to believe that prevention with the use of a vaccine is a promising strategy. At the CVD, we have pursued an approach of developing an oral, attenuated Shigella vaccine that prevents infection with the Shigella types of greatest clinical and epidemiologic importance. One of the strains to be included in the vaccine is called Shigella flexneri 2a. Investigators at the CVD have created a vaccine from Shigella flexneri 2a, designated CVD 1208S, using molecular biology techniques. To date, nearly 40 subjects have received varying doses of this vaccine with good clinical tolerance and modest immunogenicity. Previously a single dose of vaccine was used. In the current study, we will administer doses of vaccine on days 0, 28, and 56 to attempt to maximize immunogenicity. Approximately one month after the 3rd dose, a group of ~15-20 vaccinated volunteers along with a similar number of unvaccinated control subjects will be admitted to the CVD Research Isolation Ward at SNBL and challenged with wild type Shigella flexneri 2a. By comparing the attack rate of illness in vaccinated vs. unvaccinated subjects, we will determine the vaccine's ability to confer protective immunity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive
* Good general health as determined by a screening evaluation within 45 days before inoculation
* Expressed interest and availability to fulfill study requirements
* Informed, written consent
* Agrees to indefinite storage of unused clinical specimens at the CVD for use in future research, which may require separate IRB approval
* Agrees not to participate in another investigational vaccine or drug trial during the 8-month study
* Has no childbearing potential, i.e., either surgically sterilized or 1 year postmenopausal, or agrees to abstain from becoming pregnant from the day of screening (at least 14 days before vaccination) through Day 98 of the trial by using one of the following methods of birth control:

  * Abstinence;
  * Intrauterine contraceptive device;
  * Oral contraceptives or equivalent hormonal contraception, e.g., progestogen-only; implantable, cutaneous hormonal patch, injectable contraceptives, or Nuvaring (vaginal hormonal ring);
  * Diaphragm in combination with contraceptive jelly, cream, or foam;
  * Condoms with spermicide.
* Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine

Exclusion Criteria:

* An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. This includes, but is not limited to:

  * Chronic liver disease, renal insufficiency, unstable or progressive neurological disorders, diabetes mellitus, collagen vascular disease (such as lupus), active neoplastic disease (not cured or in remission), or previous hematological malignancy
  * Repeated (two or more) seizures occurring after 5 years of age, and not related to a concussion
  * Any of the following in the past 10 years: Crohn's disease, ulcerative colitis, irritable bowel disease, celiac disease, stomach or intestinal ulcers, or 2 or more episodes of arthritis (joint pain and swelling);
  * Recurrent infections (greater than 1 hospitalization for invasive bacterial infections, e.g., pneumonia, meningitis);
  * G6PD deficiency;
  * Any current illness requiring daily medication (vitamins, birth control pills, nasal or topical medications, allowed);
  * Blood in stool on more than 2 occasions (other than small amounts from straining) in past 12 months;
  * Recurrent diarrhea (greater than 5 episodes in past 6 months, each lasting 3 days or more).
* Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
* Long term (greater than 2 weeks) use of oral or parenteral steroids, or high-dose inhaled steroids (greater than 800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed)
* History of the following types of abdominal surgery:

  * Any major gastrointestinal surgery (e.g., intestinal resection or splenectomy);
  * A laparotomy for any reason (e.g., hysterectomy, Caesarian section, appendectomy, or herniorrhaphy) within the last 3 years;
  * Laparoscopic abdominal surgery within the past year.
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Known allergy or intolerance to ciprofloxacin, trimethoprim/sulfamethoxazole (or other sulfa antibiotic), ampicillin (for women), or corn
* History of shigellosis or Shigella vaccination or challenge or a laboratory worker with known exposure to Shigella
* Anticipates any of the following during the first 84 days (12 weeks) of the study:

  * Shares a household with a child less than 3 years of age, a pregnant woman or a woman who plans to become pregnant during this time;
  * Household or sexual contact with someone who has weakened immunity (such as someone with HIV infection, someone receiving treatment for cancer, or an elderly person greater than 70 years);
  * Occupation as a food-handler, childcare (for children less than 3 years), or health care worker with direct patient contact
* Poor peripheral access for placement of an intravenous line
* A clinically significant abnormality on physical examination, including, but not limited to:

  * A pathologic heart murmur
  * Lymphadenopathy
  * Hypertension (systolic blood pressure greater than 150 or diastolic blood pressure greater than 90 on 2 separate days during medical screening)
  * A large abdominal scar of unclear origin
* Any of the following laboratory abnormalities detected during medical screening:

  * WBC less than 3.0 x 103/mm3
  * Neutrophils less than 1500/mm3
  * Hemoglobin less than 12.0 g/dL (men) or less than 11.0 g/dL (women)
  * Platelets less than 130,000/mm3
  * Serum sodium less than 130 mEq/L
  * Serum creatinine greater than 1.5 mg/dL
  * SGPT greater than 82 U/L (men) or greater than 60 (women)
  * Fasting glucose greater than 99 mg/dl (if screening greater than 99 mg/dl)
  * Positive serology for syphilis, hepatitis C or HIV antibody or hepatitis B surface antigen
  * HLA B27 positive
  * Stool culture positive for Salmonella, Shigella, Campylobacter, Yersinia, Vibrio cholerae, or lacking normal flora, or pathogenic protozoa by microscopic examination.
* Positive pregnancy test during medical screening or within 24 hours of inoculation or current breast feeding (women)
* Failure to attain a score of at least 70 percent on the written examination (two attempts permitted)
* During the past 3 years, developed diarrhea during travel to a developing country, or within 1 week of returning home
* Receipt of any of the following:

  * Any vaccine or investigational drug within 30 days of study vaccine
  * A live, attenuated vaccine within the 30 days of the study vaccine
  * A subunit or killed vaccine within the 14 days of the study vaccine
  * A blood product, including immunoglobulin, in the 90 days before the study vaccine
* Receipt of antibiotics within 7 days of inoculation (or within 21 days if the antibiotic was azithromycin).
* Loose stools (grade 3-5) or any other acute illness such as fever greater than or equal to 100.0 degrees F during the 48 hours before vaccination
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant or would render the subject unable to comply with the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate, in healthy volunteers, the safety and clinical acceptability of three spaced doses (one month apart) of CVD 1208S vaccine candidate, with particular attention to the occurrence of diarrhea, dysentery, and fever | approximately June 2009-January 2010 and October 2010
To characterize the following immune responses following ingestion of this vaccine: Serum IgA and IgG anti-S. flexneri 2a lipopolysaccharide (LPS) antibody and IgA anti-LPS antibody secreting cells (ASC) | approximately June 2009, February 2010 - April 2010, and October 2010

SECONDARY OUTCOMES:
To assess the fecal shedding of CVD 1208S | approximately June - July 2009 and October 2010
To elucidate the systemic and mucosal immune responses to vaccination, including fecal IgA antibodies to LPS and Ipas, IgG anti-LPS ASCs, IgG and IgA Ipa ASC, ASC & T cell homing, specific B and T memory responses, and cytokine production by PBMC. | approximately June 2009 and August - October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Kotloff, M.D., Principal Investigator — University of Maryland, Baltimore Center for Vaccine Development
Locations (1):
- University of Maryland, Baltimore Center for Vaccine Development, Baltimore, Maryland, United States